CLINICAL TRIAL: NCT04882761
Title: Evaluation of Soft Tissue Stability and Labial Plate of Bone of Immediate Implant in Direct Contact Versus Gap With Socket Shield (A Randomized Clinical Study)
Brief Title: Socket Shield With Immediate Implant Stability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13875
Record Dates: First submitted 2021-02-27; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Dental Implant
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Socket shield in direct contact with dental implant (Active Comparator): eight partially extracted sockets where implant (Neobiotech) was placed in direct contact to socket shield
  Interventions: Device: Dental implant
- Socket shield with gap and xenograft with dental implant (Active Comparator): eight partially extracted sockets where a gap was left between implant (Neobiotech) and socket shield
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — Comparative

SUMMARY:
To evaluate socket shield technique either placing implant in direct contact to tooth fragment versus gap created between the tooth and implant.

DETAILED DESCRIPTION:
Patients with a non-restorable tooth located in anterior maxillary arch was included in this study, patients were divided into two groups, eight implants per group, both groups had socket shield, group 1 will have implant in direct contact with shield, second group had a gap between dental implant and shield. soft tissue stability, bone width and implant stability was assessed preoperatively, immediate and 6 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a non-restorable tooth located in anterior maxillary arch (upper right second premolar to upper left second premolar). Tooth to be extracted is endodontically treated and free from periapical infection.
2. Systemic free patients according to modified Cornell medical index (Brodmank and Erdmann 1949).
3. Patients with good compliance.

Exclusion Criteria:

1. Teeth with current acute periapical infection or sinus tracts.
2. Heavy smokers and patients with bruxism habits.
3. Patients with poor oral hygiene or not willing to perform oral hygiene measures.
4. Vulnerable groups (as pregnant females and decisionally impaired individuals).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Soft tissue stability | 6 months postoperatively
  Pink esthetic score

SECONDARY OUTCOMES:
Bone stability | 6 months postoperatively
  By Ostell

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Adel-Khattab, PhD, Study Director — Ain Shams University
Locations (1):
- Doaa Khattab, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No